CLINICAL TRIAL: NCT06853990
Title: A Single-arm Trial With an Innovative Automated Insulin Delivery System for Type 2 Diabetes ("Twiist-T2D")
Brief Title: Innovative Automated Insulin Delivery System for Type 2 Diabetes
Acronym: twiist-T2D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deka Research and Development (Industry)
Collaborators: Sequel Med Tech (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DKPI-00730-001
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Insulin Treated Type 2 Diabetes Mellitus
Keywords: automated insulin delivery system (AID)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- twiist users (Experimental)
  Interventions: Device: twiist insulin delivery system

INTERVENTIONS:
Device: twiist insulin delivery system — twiist system includes a novel insulin pump, a CGM sensor and the DEKA Loop algorithm

SUMMARY:
The goal of this clinical trial is to learn if the twiist insulin delivery system works to treat adults with insulin-treated type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old at the time of screening (date informed consent form signed)
2. Clinical diagnosis of type 2 diabetes based on investigator assessment of at least 6 months duration at time of screening.
3. Using one of the following insulin regimens for at least 13 weeks prior to screening: (1) basal-bolus insulin therapy with at least one injection containing rapid-acting insulin per day, (2) open-loop insulin pump, (3) premixed insulin with a rapid component, (4) basal insulin without bolus insulin.
4. If using noninsulin glucose-lowering medications (such as GLP-1 receptor agonist, SGLT2 inhibitor, or other) or weight-reduction medications that can have a meaningful effect on glycemia, dose has been stable for at least 4 weeks prior to screening in the judgement of the investigator, and there are no plans to change the dose during the duration of the study. If not using glucose-lowering or weight-reduction medications that can have a meaningful effect on glycemia, participant agrees to not initiate such medications during the duration of the study.
5. Willing and able to use only insulin approved for use in the study pump.
6. Has the ability to read and understand written English or another language available as an option for the pump's user interface.
7. Investigator believes that the participant has the cognitive capacity to provide informed consent.
8. Investigator believes that the participant can successfully and safely operate all study devices and is capable of adhering to the protocol and completing the study.

   a. This includes considering the potential impact of medical conditions known to be present including cardiovascular, liver, kidney disease, thyroid disease, adrenal disease, malignancies, vision difficulties, active proliferative retinopathy, and other medical conditions; psychiatric conditions including eating disorders; drug or alcohol abuse.
9. Willing to participate in the study meal and exercise challenges and have a care partner willing to be trained in hypoglycemia treatment guidelines present during and immediately after the exercise challenges (not required if exercise sessions will be done in clinic).
10. Participants capable of becoming pregnant must meet one of the following criteria:

    a. Has a negative urine pregnancy test and agrees to use one of the accepted contraceptive regimens throughout the entire duration of the trial from screening until last follow-up visit. The following contraceptive measures are considered adequate: i. Combined estrogen and progesterone containing hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal).

ii. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable).

iii. Placement of an intrauterine device or intrauterine hormone-releasing system.

iv. Bilateral tubal occlusion. v. Barrier methods of contraception (condom or occlusive cap with spermicidal foam/gel/film/cream/suppository).

vi. Has a vasectomized or sterile partner (where partner is sole partner of subject) and where vasectomy has been confirmed by medical assessment.

vii. Exercises true sexual abstinence. Sexual abstinence is defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.

or b. Participant is of non-childbearing potential due to menopause with at least one year since last menses or a medical condition confirmed by the investigator.

Exclusion Criteria:

1. Type 1 diabetes
2. Use of an FDA-approved or non-FDA approved closed-loop or hybrid closed-loop insulin delivery system within the past 3 months.
3. Pregnancy (as demonstrated by a positive test) or breast-feeding at time of screening or planning to become pregnant during the next 4 months.
4. Concomitant disease or condition that in the opinion of the investigator may compromise patient safety including but not limited to; cystic fibrosis, severe mental illness, a diagnosed or suspected eating disorder or any uncontrolled long term medical condition that would interfere with study related tasks or visits.
5. Current use of implantable CGM sensor (e.g., Senseonics)
6. Current use of at least 500 mg of ascorbic acid (Vitamin C)
7. Presence of a hemoglobinopathy or other condition that is expected to affect the measurement of HbA1c in the judgment of the investigator.
8. Immediate family member (spouse, child, sibling, parent) of any person at an investigative site who is directly affiliated with this study or who is an employee of Sequel Med Tech, Millyard Advanced Medical Products LLC, Merrimack Manufacturing, or DEKA Research and Development Corp.
9. More than 2 severe hypoglycemic events requiring third party help or hospitalization within the last 6 months prior to screening
10. More than one DKA or HHS event within the last 6 months prior to screening
11. Lack of reliable telephone or internet service (for contact)
12. Known allergy to medical grade adhesives or skin condition that precludes use of the study pump or CGM
13. Current participation in another diabetes-related interventional clinical trial.
14. Anticipated change of residency or travel for more than 14 days at a time during the study that may, per investigator judgment, interfere with the completion of study visits, contacts, or procedures.
15. Feasibility Phase only: Clarke Hypoglycemia Awareness Survey score of 4 or greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline to 13-weeks
  HbA1c will be tested first for non-inferiority (non-inferiority limit 0.3%) and then if non-inferiority is demonstrated, it will be tested for superiority.

SECONDARY OUTCOMES:
CGM-measured time in and out of range | Baseline to 13-weeks
  For the following endpoints, the change from baseline to follow-up will be tested in a hierarchy to control the overall type 1 error (assuming the analysis of the primary endpoint is statistically significant). Testing will be for superiority unless otherwise specified.
  * CGM-measured time in range 70-180 mg/dL
  * CGM-measured time in tight range 70-140 mg/dL
  * CGM-measured time <54 mg/dL (non-inferiority, margin 0.5%)
  * CGM-measured time <70 mg/dL (non-inferiority, margin 2.0%)
  * CGM-measured mean glucose
  * CGM-measured time >180 mg/dL
  * CGM-measured time >250 mg/dL
  * CGM-measured time <70 mg/dL
  * CGM-measured time <54 mg/dL

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - University of Colorado, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Endocrine Research Solutions, Inc, Roswell, Georgia
  - Rocky Mountain Clinical Research, LLC, Idaho Falls, Idaho
  - Endeavor Health, Skokie, Illinois
  - IU Health University Hospital, Indianapolis, Indiana
  - Iowa Diabetes & Endocrinology Research Center, West Des Moines, Iowa
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health, Detroit, Michigan
  - International Diabetes Center - Health Partners Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Naomi Berrie Diabetes Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Diabetes & Endocrine Treatment Specialists, Sandy City, Utah
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No